CLINICAL TRIAL: NCT05304845
Title: A Randomized, Open-label Study to Evaluate the Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of Drug-drug Interactions Between DWP14012 and Aspirin in Healthy Subjects
Brief Title: Drug-drug Interactions Between DWP14012 and Aspirin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DW_DWP14012108
Record Dates: First submitted 2022-03-16; First posted 2022-03-31 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-03

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — fexuprazan; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Aspirin (substrate), DWP14012 (Perpetrator)
  Interventions: Drug: DWP14012; Drug: Aspirin
- Cohort 2 (Experimental): DWP14012 (substrate), Aspirin (Perpetrator)
  Interventions: Drug: DWP14012; Drug: Aspirin

INTERVENTIONS:
Drug: DWP14012 — Potassium-competitive acid blocker
Drug: Aspirin — acetylsalicylic acid

SUMMARY:
This is a randomized, open-label study to evaluate the safety/tolerability and PK/PD drug-drug interactions between DWP14012 and aspirin when administered in combination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 and ≤ 50 years at screening
* Subjects with a body weight ≥ 50.0 kg to ≤ 90.0 kg with a body mass index (BMI) of ≥ 18.0 kg/m2 to ≤ 27.0 kg/m2 at screening

  ※ BMI (kg/m2) = body weight (kg)/[height (m)]2
* Subjects who voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a sufficient explanation on this study and fully understanding the information
* Subjects who are eligible to participate in the study at the discretion of the investigator by physical examination, laboratory tests, and investigator questioning, etc.
* For women, negative urine pregnancy test (hCG) at the screening visit

Exclusion Criteria:

* Subjects with hypersensitivity or history of clinically significant hypersensitivity to drugs including potassium competitive acid blocker [P-CAB] class, aspirin, salicylic acid, or other drugs (non-steroidal anti-inflammatory drug [NSAIDs], antibiotics, etc.)
* Women who are or may be pregnant, or are breast-feeding
* Subjects with a history related to blood clotting disorder or bleeding
* Subjects with a medical diagnosis of functional constipation
* Subjects with a history of drug abuse or a positive result of using abusive drugs in the urine drug screen
* Subjects who participated in other clinical trials (including bioequivalence studies) within 6 months prior to the first scheduled dose of the IP
* Subjects who donated whole blood within 2 months, donated blood components within 1 month, or received blood transfusion within 1 month prior to the first scheduled dose
* Subjects who are unable to refrain from grapefruit-containing products from 3 days prior to the first scheduled dose until last discharge from hospital
* Subjects or their spouses or partners who are unable to use medically acceptable appropriate double-method of contraception or medically acceptable contraception throughout the study period and for at least 4 weeks after the last IP administration, and disagreed to refrain from donating sperms during this period
* Subjects with hereditary disorders including galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Cmax of aspirin | Up to 21 days
Cmax,ss of DWP14012 | Up to 13 days
Emax | Up to 21 days
AUClast of aspirin | Up to 21 days
AUCτ,ss of DWP14012 | Up to 13 days
time to Emax | Up to 21 days
AUEC | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: In Jin Jang, MD, PhD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No